CLINICAL TRIAL: NCT02646709
Title: The Effect of Different Doses of Ketamine on Tracheal Intubating Conditions Using Low Dose Rocuronium in Children
Brief Title: The Effect of Different Dose of Ketamine With Low Dose Rocuronium in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Go Un Roh, principal investigator, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: AJIRB-MED-CT4-15-153
Record Dates: First submitted 2015-12-28; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ketamine 1 (Experimental): Ketamine 1 mg/kg will be injected during induction. Low dose rocuronium (0.3 mg/kg) will be injected for muscle relaxation.
  Interventions: Drug: Rocuronium; Drug: ketamine 1
- Ketamine 1.5 (Experimental): Ketamine 1.5 mg/kg will be injected during induction. Low dose rocuronium (0.3 mg/kg) will be injected for muscle relaxation.
  Interventions: Drug: Rocuronium; Drug: ketamine 1.5
- Ketamine 2 (Experimental): Ketamine 2 mg/kg will be injected during induction. Low dose rocuronium (0.3 mg/kg) will be injected for muscle relaxation.
  Interventions: Drug: Rocuronium; Drug: ketamine 2

INTERVENTIONS:
Drug: Rocuronium — Low dose rocuronium (0.3 mg/kg) will be injected after induction of anesthesia with ketamine.
Drug: ketamine 1 — ketamine 1 mg/kg will be injected for induction of anesthesia
  Arms: Ketamine 1
Drug: ketamine 1.5 — ketamine 1.5 mg/kg will be injected for induction of anesthesia
  Arms: Ketamine 1.5
Drug: ketamine 2 — ketamine 2 mg/kg will be injected for induction of anesthesia
  Arms: Ketamine 2

SUMMARY:
Rocuronium is suitable for rapid induction within 60-90 seconds and its effect last 24-40 minute after single bolus injection. For outpatient surgery with short operation time, low dose rocuronium is frequently used for rapid recovery at the expense of compromised intubating condition. For better intubating condition, ketamine can be used. However, appropriate dose of ketamine with low dose rocuronium is not established yet. This study, 3 different doses of ketamine with low dose rocuronium will be compared for appropriate intubating condition.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I, II

Exclusion Criteria:

* upper respiratory infection within 14 days
* anticipated difficult intubation

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Intubation Condition | during and after intubation, about 2 minute
  5 variables will be individually evaluated though 3 point scale (excellent, good, poor). If all variables are graded as excellent, intubation condition will be excellent. If at least 1 variable is poor, it will be reported as poor. Otherwise, it will be reported as good.
  1. Laryngoscope easiness
  2. Vocal cord position
  3. Vocal cord movement
  4. Movement of limb
  5. Coughing

SECONDARY OUTCOMES:
heart rate | 1. 1 min before induction 2.1 min after ketamine injection 3. 1min after intubation 4. 5 min after intubation 5. 10 min after intubation
  heart rate will be recorded.
time for extubation | from the end of surgery to extubation, within 10 min
emergence agitation (4 points scale) | 5 min after postanesthesia care unit (PACU) admission
  4 points scale
  1: calm 2. cry but manageable 3. cry, not manageable 4. excitation
PACU time | from PACU admission to discharge, about 30 min
severity of vomiting | 1. 1 min after PACU admission 2. 30 min after PACU admission
  severity(0-10)
Analgesic requirements (mg/kg) | during PACU stay, about 30 min
  if pain score exceed 3, fentanyl will be introduced. The total dose of fentanyl injection will be recorded.
Desaturation | during PACU stay, about 30 min
  pulseoximeter will be applied and peripheral oxygen saturation less than 94 will be recorded.
blood pressure | 1. 1 min before induction 2.1 min after ketamine injection 3. 1min after intubation 4. 5 min after intubation 5. 10 min after intubation
  blood pressure will be recorded
frequency of vomiting | 1. 1 min after PACU admission 2. 30 min after PACU admission

CONTACTS AND LOCATIONS:
Overall Officials: Go Un Roh, MD, Principal Investigator — Ajou University School of Medicine

IPD SHARING:
Plan to Share IPD: No